CLINICAL TRIAL: NCT01155401
Title: Study of Incidence of Drug-induced Upper Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GRU-NEX-2009/2
Record Dates: First submitted 2010-06-25; First posted 2010-07-01 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: acute upper gastrointestinal bleeding; patients with drug-induced upper gastrointestinal bleeding; routine management
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with acute upper gastrointestinal bleeding

SUMMARY:
The purpose of this study is to determine and analyse the incidence, severity, risk factors and routine management of acute drug-induced upper gastrointestinal bleeding (UGIB) in the population of Russian patients

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of acute upper gastrointestinal bleeding, confirmed by presence of hematemesis/ coffee ground vomiting, melena, as well as other clinical or laboratory evidence of acute blood loss from the upper gastrointestinal tract
* Written informed consent provided prior the start of participation in the study.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with drug-induced upper gastrointestinal bleeding | About 1 year

SECONDARY OUTCOMES:
Number and percentage of patients with each symptom and each Forrest class of upper gastrointestinal bleeding | About 1 year
Number and percentage of patients with concomitant diseases contributing to drug-induced upper gastrointestinal bleeding and those who receive NSAIDs, antiplatelet agents, anticoagulants, steroids or combination therapy | About 1 year
Number and percentage of patients with each type of bleeding outcomes who received different types of hemostatic therapy | About 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Boris R Gelfand, Prof, Principal Investigator — Department of the Russian State Medical University
Locations (1):
- Research Site, Moscow, Russia